CLINICAL TRIAL: NCT06235489
Title: "Evaluation of Clinical Performance of a Flowable Bulk Fill Composite Resin Versus a Highly Viscous Glass Ionomer Cement in Class II Cavities in Primary Molars: A Randomized Clinical Trial"
Brief Title: Evaluation of Clinical Success of Bulk Fil Composite Versus Highly Viscous Glass Ionomer in Primary Class II Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Abdel Azim, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PED 22-5D
Record Dates: First submitted 2023-11-22; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Dental Caries Class II
Keywords: HVGIC; Proximal caries; Bulk-fil flowable composite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palfique Bulk Flow bulk-fil flowable restorative material (Experimental): Procedure: restoration of proximal cavities of primary molars with bulk-fil flowable composite removal of proximal caries of primary molars and restoration of the cavities prepared by Palfique bulk flow
  Interventions: Other: Palfique Bulk Flow
- Glass-hybrid added HVGIC Equia Forte HT Glass-hyrbid-added highly viscous glass ionomer cement (Active Comparator): Procedure: Restoration of proximal cavities of primary molars with highly viscous glass ionomer cement removal of proximal caries of primary molars and restoration of the cavities prepared by the Equia forte HT
  Interventions: Other: Palfique Bulk Flow

INTERVENTIONS:
Other: Palfique Bulk Flow — removal of caries in primary molars and placement of restorative materials
  Other Names: Equia Forte HT

SUMMARY:
evaluate the clinical performance of EQUIA Forte ® ( a HVGIC) and Plafique® Bulk Flow composite resin when placed in class II cavities in primary molars.

DETAILED DESCRIPTION:
1. Thorough diagnosis of patients will be done by the primary investigator. Patients with class II carious primary molars with score 4 or 5 using the International Caries Detections and Assessment Criteria (ICDAS).
2. Pre-operative bitewing radiographs will be obtained to assess the depth of the cavity. Primary molars with score D1 or D2 according to the ADA will be included in the study.
3. Each patient will be assigned to one of the two groups.

   * Group I (n= 59): Plafique Bulk Flow Composite.
   * Group II (n=59): EQUIA Forte Group.
4. Class II carious primary molars are prepared using 330 burs. The cavity will be approximately with a depth of 0.5 mm in dentin and width of at least one-third of the occlusal table. Outline of the cavity will be determined by the extent of the carious lesion. No beveling will be done in any of the cavities.
5. Matrix is placed and secured in position.
6. One of the 2 restorative materials is placed in the cavity using the manufacturer's instructions.
7. Patients will be recalled at 3, 6, and 12 months to evaluate the restoration clinically using the FDI criteria.
8. Patients will receive oral health education on how to maintain a proper oral hygiene and proper diet consumption.
9. They will be given manual tooth brushes and tooth pastes to use during the study.

ELIGIBILITY:
Inclusion Criteria:

* Four to 8 years old children
* Cooperative children classified as class 3 or 4 based on Frankle et al. classification.
* Presence of deep bite or any type of malocclusion or parafunctional habits.
* Children who have at least one primary molar with active proximal caries (score 4 or 5 using ICDAS).

Exclusion Criteria:

* Refusal of the parents to sign the informed consent.
* Presence of deep bite or any type of malocclusion or parafunctional habits.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
clinical performance | one- year
  Evaluate and compare the clinical performance of two commercially available bulk restorative materials (Plafique® Bulk Flow Composite and EQUIA Forte®) for 12 months using the Federation Dentaire Internationale (FDI) criteria when placed in class II cavity in primary molars.
  This diagnostic system classified aesthetic, functional, and biological properties and covers various types of failures by using 16 different categories with five grades for each criterion.
  Where score 1 indicates clinically excellent/very good (sufficient), 2: clinically good (sufficient), 3: Clinically satisfactory (sufficient), 4: Clinically unsatisfactory (partially insufficient), and finally score 5 indicates clinically poor (entirely insufficient)

CONTACTS AND LOCATIONS:
Overall Officials: Mariem O Wassel, Prof, Study Director — Head of Pediatric Dentistry Department, Faculty of Dentistry, Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No